CLINICAL TRIAL: NCT05027204
Title: A Single-arm, Multicenter, Phase Ib/II Clinical Study of Docetaxel for Injection (Albumin-bound) in Combination With Nivolumab in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN) Progressing on or After Platinum-based Therapy
Brief Title: A Study of Docetaxel for Injection (Albumin-bound) in Combination With Nivolumab in Patients With Head and Neck (SCCHN)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HB1801-CSP-003
Record Dates: First submitted 2021-08-19; First posted 2021-08-30 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-01

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Docetaxel; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Docetaxel combined with Nivolumab (Experimental): Phase Ib: The eligible patients with SCCHN will received Docetaxel for Injection (Albumin-bound) 75 mg/m^2 or 100 mg/m^2 sequentially in combination with Nivolumab 360 mg to evaluate safety and efficacy and explore RP2D.
  Phase II: According to the RP2D determined in the phase Ib study, patients will be treated with Docetaxel for Injection (Albumin-bound) combined with Nivolumab until participants meet the criteria for termination or withdrawal criteria, for a maximum of 2 years.
  Interventions: Drug: Docetaxel; Drug: Nivolumab

INTERVENTIONS:
Drug: Docetaxel — Docetaxel for Injection (Albumin-bound), Q3W, i.v. 60 min
Drug: Nivolumab — Nivolumab, Q3W, i.v. 30 min

SUMMARY:
This trial is a single-arm, multicenter phase Ib/II clinical study to evaluate the efficacy and safety of Docetaxel for Injection (Albumin-bound) combined with Nivolumab and the pharmacokinetic characteristics of Docetaxel in patients with recurrent or metastatic SCCHN who are positive for PD-L1 expression and have progressed on or after platinum-based therapy.

DETAILED DESCRIPTION:
This study will be conducted in two stages (phase Ib and phase II). Phase Ib: To explore the safety and tolerability of Docetaxel for Injection (Albumin-bound) (75 mg/m^2 and 100 mg/m^2) combined with Nivolumab 360 mg. Dose exploration will be started at low dose and proceed in turn.

Phase II: According to the recommended phase II dose (RP2D) determined in the phase Ib study, a phase II study of Docetaxel for Injection (Albumin-bound) combined with Nivolumab will be conducted to observe the efficacy of the combination regimen, with ORR as the primary study endpoint. Simon's optimal 2-stage design will be adopted for phase II study.

All patients in Phase Ib and Phase II will be treated with Docetaxel for Injection (Albumin-bound) combined with Nivolumab until participants meet the criteria for termination or withdrawal criteria, for a maximum of 2 years

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old and voluntarily signed the informed consent form.
2. Patients with histologically or cytologically confirmed SCCHN (primary tumor located in the oral cavity, oropharynx, larynx or hypopharynx), with positive PD-L1 expression, and who are not suitable for local radical therapy.
3. Patients with platinum-based regimen failure, defined as:

   1. . Recurrent or metastatic SCCHN with disease progression during or after platinum-based therapy;
   2. . Locally advanced head and neck carcinoma with recurrence or metastasis within 6 months after platinum-based therapy in previous multimodal therapy.
4. Previous or qualified tumor tissue samples are available for testing PD-L1.
5. Patients with oropharyngeal carcinoma should provide previous HPVp16 immunohistochemical test results, or eligible tumor tissue samples for testing HPV status.
6. At least one measurable lesion confirmed by CT or MRI according to RECISTv1.1 (previously irradiated, progressive disease or tumor persistence ≥ 3 months after radiotherapy can be considered as measurable lesions).
7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
8. Life expectancy ≥ 3 months.
9. Main organ function meets the following criteria within 7 days before treatment (no medical supportive treatments such as blood component transfusion, human granulocyte colony-stimulating factor (G-CSF), thrombopoietin (TPO), interleukin-11, and erythropoietin (EPO) within 2 weeks before administration of the investigational product).

   Absolute neutrophil count ≥1.5×10^9/L Platelets ≥90×10^9/L Hb≥90 g/L or ≥5.6 mmol/L Serum creatinine ≤ 1.5×ULN or creatinine clearance rate ≥ 40 mL/min Total bilirubin ≤1.0×ULN (≤ 1.5 × ULN for patients with liver metastasis or liver cancer); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 × ULN ( ≤ 2.5 × ULN for patients with liver metastasis or liver cancer); Activated Partial Thromboplastin Time (APTT) ≤ 1.5×ULN, International Normalized Ratio (INR) ≤ 1.5×ULN.
10. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days prior to the first dose of the investigational drug. The patient and his/her spouse must agree to take adequate contraception from signing of ICF through 6 months after last dose, during which time women should be nonlactating and men should refrain from donating sperm.

Exclusion Criteria:

1. Histologically or cytologically confirmed recurrent or metastatic nasopharyngeal carcinoma, SCCHN with unknown primary lesion, salivary gland carcinoma, or non-squamous tissue carcinoma (e.g., mucosal melanoma).
2. Patients with active brain metastasis and leptomeningeal metastasis. Patients with brain metastasis for whom there is no evidence of PD by MRI at least 8 weeks after treatment and within 28 days before the first dose of the investigational drug can be included; Those who do not require systemic cortisol therapy (prednisone > 10 mg/day or equivalent) at least 2 weeks before the first dose of the investigational drug can be included; Patients with skull base lesions without definite evidence of dural or parenchymal brain involvement can be considered to be included only after discussion with the sponsor's medical monitor.
3. History of other malignancies within 5 years prior to the first dose of the investigational drug, except for the following: a. Any other invasive malignancy (for which the patient has received adequate treatment) with disease free status lasting > 3 years, which will not affect the assessment of tumor efficacy as assessed by the investigator; b. Cured basal cell or squamous cell skin carcinoma, superficial bladder cancer, prostate cancer, cervical cancer, or breast cancer in situ, and other locally curable cancers.
4. Patients with known or suspected autoimmune disease within 2 years before the first dose of the investigational drug, except for the following: a. well-controlled type I diabetes; b. well-controlled hypothyroidism requiring only hormone replacement therapy; c. skin diseases (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment; d. patients who are not expected to relapse in the absence of external triggers.
5. Patients with an uncontrollable third space effusion (e.g. pleural effusion, ascites, or pericardial effusion), who, in the judgment of the investigator, are not suitable for the study.
6. Patients with a history of severe cardiovascular disease within 6 months before the first dose of the investigational drug, including but not limited to:

   1. . Severe heart rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention and third-degree atrioventricular block;
   2. . History of myocardial infarction, angina pectoris, angioplasty and coronary artery bypass surgery;
   3. . Heart failure with New York Heart Association (NYHA) Classification of Class III and above;
   4. . Poorly controlled hypertension.
7. Patients with prolonged QT/QTc interval (QTcF > 480 ms, Fridericia's formula: QTcF = QT/RR^0.33, RR = 60/heart rate) by ECG during the screening period and/or with left ventricular ejection fraction (LVEF) ≤ 50% by echocardiography (ECHO) or multi-gated acquisition (MUGA) during the screening period;
8. Patients with positive HCV antibody (+) (patients with negative HCV RNA can be included, and anti-HCV treatment other than interferon is allowed), active hepatitis B (patients with HBV DNA ≤ 500 IU/mL can be included, and anti-HBV treatment other than interferon is allowed), known HIV positive or known acquired immunodeficiency syndrome (AIDS) during the screening period.
9. Patients who have undergone major organ surgery within 4 weeks before the first dose of the investigational drug, or who need to undergo elective surgery during the study.
10. Patients who fail to recover from the toxic responses caused by previous anti-tumor treatment to Grade 1 and below (CTCAE 5.0), except for the following: Grade 2 neuropathy, alopecia, hypothyroidism caused by previous anti-tumor treatment (including hormone replacement therapy) and toxicity without safety risks as judged by the investigator.
11. Patients who have previously received T cell costimulating drugs or drugs acting on immune checkpoint pathways (including PD-1, PD-L1/2, CTLA-4 inhibitors, etc.).
12. Patients who have previously received other immunotherapies and experienced ≥ Grade 3 irAE (immune-related adverse event).
13. Patients who have previously received taxanes (patients who previously received taxane-containing induction chemotherapy and progressed after 6 months can be included).
14. Patients who have received anti-tumor treatments such as chemotherapy, radiotherapy, targeted therapy, immunotherapy and other clinical study drugs within 4 weeks before the first dose of the investigational drug, and other conditions are as follows:

    Local palliative radiotherapy within 2 weeks before the first dose of the investigational drug; oral fluoropyrimidines, small molecule targeted drugs, etc. within 2 weeks before the first dose of the investigational drug or within known 5 half-lives of the drug (whichever is longer); Traditional Chinese medicines with anti-tumor indications within 2 weeks before the first dose of the investigational drug.
15. Patients who have received corticosteroid (prednisone > 10 mg/day or equivalent) or other immunosuppressive therapies within 2 weeks before the first dose of the investigational drug, except for the following: a. use of topical, ocular, intra-articular, intranasal and inhaled glucocorticoids; b. short-term use of glucocorticoids for prophylaxis (such as prevention of contrast agent allergy).
16. Patients who have received live attenuated vaccine within 2 weeks before the first dose of the investigational drug or planned to receive live attenuated vaccine during the study period.
17. Patients who have used potent inhibitors or inducers of CYP3A4 within 2 weeks before the first dose of the investigational drug.
18. Patients with known ≥ Grade 3 hypersensitivity and/or contraindication to albumin or monoclonal antibodies.
19. Other situations that the investigator considers not suitable for participating in the clinical study, including but not limited to: the patient is complicated by severe or uncontrolled medical conditions, which interfere with the interpretation of study results and affect the study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2022-03-04 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Incidence of adverse events and serious adverse events | 6 weeks
  Incidence of adverse events and serious adverse events
Phase II: Objective response rate (ORR) | 2 years
  Objective response rate

SECONDARY OUTCOMES:
The pharmacokinetic parameters (free docetaxel and total docetaxel) : AUC0-last | 24 hours
  Area under the plasma concentration versus time curve (AUC)
The pharmacokinetic parameters (free docetaxel and total docetaxel) : AUC0-∞ | 24 hours
  Area under the plasma concentration versus time curve (AUC)
The pharmacokinetic parameters (free docetaxel and total docetaxel) : Cmax | 24 hours
  The Cmax is the maximum observed serum concentration of Docetaxel
The pharmacokinetic parameters (free docetaxel and total docetaxel) : Tmax | 24 hours
  The Tmax is the time at which the maximum concentration of Docetaxel
The pharmacokinetic parameters (free docetaxel and total docetaxel) : t½ | 24 hours
  Terminal elimination half-life (t1/2) of docetaxel
The pharmacokinetic parameters (free docetaxel and total docetaxel) : Vd | 24 hours
  Volume of distribtion of docetaxel
The pharmacokinetic parameters (free docetaxel and total docetaxel) : CL | 24 hours
  Clearance of Docetaxel
Phase II: Disease control rate (DCR) | 2 years
  Disease control rate
Phase II: Duration of response (DOR) | 2 years
  Duration of response
Phase II: Progression-free survival (PFS) | 2 years
  Progression-free survival
Phase II: Overall survival (OS) | 2 years
  Overall survival
Phase II: Incidence of adverse events and serious adverse events | 2 years
  Incidence of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Guo Ye, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No